CLINICAL TRIAL: NCT02340546
Title: Trajectory Changes of Coronary Sinus Lead Tip and Cardiac Resynchronization Therapy Outcome
Acronym: TRAJECTORIES
Status: Completed | Type: Observational
Sponsor: Corrado Tomasi (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor-Investigator, Corrado Tomasi, Cardiologist, Chief Electrophisiologist of the Cardiovascular Department, Ospedale Santa Maria delle Croci
Organization: Ospedale Santa Maria delle Croci (Other)
Other Study IDs: 1368/2014
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure; Left-Sided Heart Failure; Ventricular Dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: cardiac resynchronization therapy — cardiac resynchronization by means of biventricular pacing via left ventricular pace from coronary sinus veins combined with conventional any-site right ventricular pace

SUMMARY:
In chronic systolic heart failure patients submitted to cardiac resynchronization therapy, the study aims at assessing whether geometric variations in coronary sinus lead tip trajectory throughout the cardiac cycle acutely induced by biventricular pacing, are predictive of the volumetric and clinical response to the treatment at six-month follow-up.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) has become a standard treatment in patients with symptomatic chronic systolic heart failure, reduced left ventricular (LV) function and wide electrocardiographic ventricular (QRS) complex, but approximately one third of patients do not respond to the treatment. Current ability to predict long-term response to CRT at implant is slight. Investigations have focused mostly on early prediction of the reversal of LV remodeling by means of LV pacing, which is delivered more frequently as biventricular pacing, combined with conventional right ventricular (RV) pacing. LV dyssynchrony areas have been identified as suitable targets for pacing, but no methods still can evaluate real-time, intra-operative acute effects of pacing on LV mechanics. This issue has become even more evident in the subset of CS implants of quadripolar leads, which offer relevant advantages but highlight the lack of methods for selecting the pacing configuration among the safe and effective ones.

Since LV pacing is currently delivered on the epicardium by a lead inserted in coronary sinus (CS) branches, the interface between the point of pacing delivery on LV surface and the underlying LV wall, and overall lead movements inside coronary sinus might describe some underlying myocardial mechanics. By means of a recently published fluoroscopy-based method, the trajectory of the electrode tip inserted in CS branches can be reconstructed in three-dimensions (3D) throughout the cardiac cycle. A preliminary clinical pilot study (Heart Rhythm 2013;10:1360) demonstrated that biventricular pacing acutely induced changes in trajectory geometry, which were correlated to the echocardiographic volumetric response to CRT at six-month post-implant follow-up. In responders only, biventricular pace abruptly determined a more circular shape. Such results were "hypothesis-generating" and are to be yet tested on a larger scale.

The study analyzes the predictive power of the changes in pacing cathode trajectory metrics occurring at the start of biventricular pacing with respect to both:

1. the volumetric response to CRT, measured at six-month follow-up by a unique criterion;
2. the clinical response to CRT, described at six-month follow-up by three clinical indices.

Secondarily, this study evaluates whether trajectory variations would be able to acutely guide the selection of the definitive LV pacing configuration in the subset of implants of a CS quadripolar lead.

The trajectory geometry metrics to analyze are:

* trajectory length;
* area of the surface encompassed by the trajectory in the 3D space;
* trajectory mean curvature;
* the three singular values indicating to what extent the trajectory is distributed along each of its three principal directions (eigenvectors);
* ratio between the two main singular values, indicating to what extent the trajectory is distributed along only one (principal) direction;
* trajectory eccentricity;
* distance between the trajectory barycenter.

Operatively:

* patients submitted to implant of a CRT device (pacemaker or implantable cardioverter defibrillator) according to current indications are evaluated;
* all market-released CRT devices can be implanted; the choice of CS lead, implantation technique, leads placement is left to each investigator decision;
* during implant procedure, the devices are programmed in sense-only mode; if upgrades, the pre-existing pacing programming is kept unmodified until the start of biventricular stimulation;
* short fluoroscopy recordings of lead movements inside CS branching are taken in three radiological projections (posteroanterior, 30° right and left anterior oblique), both just before and immediately after the beginning of biventricular pacing at prefixed settings, which are: lower rate at 60-70 beats per min; atrioventricular (AV) delay at 120 ms and interventricular (VV) delay at 0 ms;
* in the subset of implants of a quadripolar lead, other two fluoroscopic recordings are acutely acquired during a short period of pacing from each of two other cathodes, which are predefined as being at 20-35 mm and 40-50 mm from lead tip;
* 3D trajectories are reconstructed for the lead tip (the distal pole), and, in quadripolar lead implants, also for other two pacing cathodes, both before and acutely at biventricular pacing start;
* after acquisition, at any time pacing settings can be optimized and modified at investigators choice;
* if a quadripolar CS lead is used, the pacing configuration at discharge is preferably chosen as that associated with the largest change of cathode trajectory towards a more circular shape at biventricular pace start;
* CRT device checking is scheduled at 6-month follow-up; other checks are left to the discretion of each center; a visit is advised at 30-60 days after discharge;
* all centers arrange for the two index echocardiographic evaluations to be performed on schedule by an expert operator, who has to be blinded about any trajectory results, and according to recommendations of the American Society of Echocardiography. All examinations are recorded on external support (analogic or digital) and handed to the internal Echocardiography Core-Lab, which is identified among participating institutions. The Echo Core-Lab operator(s) is not directly involved in the study and is kept unaware of all trajectory results up to the end of the study;
* the fluoroscopic recordings are stored on a CD and analyzed off-line by the Engineering Core Lab, using the method previously published.

The following variables are collected at baseline

- age, gender, height and weight; presence of diabetes, hypertension, chronic obstructive bronchopneumopathy, previous stroke, previous myocardial infarction; moderate to severe valvular heart disease; any previous myocardial revascularization; previous heart surgery; chronic renal failure,defined by glomerular filtration rate (eGFR) <60 mL/min/1.73 square metre; current value of eGFR (mL/min/1.73 square metre); current medical treatment with beta-blockers, diuretics, ACE inhibitors, angiotensin II antagonists, aldosterone antagonists, antiarrhythmic, oral anticoagulants, anti-platelets.

The following variables are collected both at peri-implant and at six-month follow-up:

1. Clinical : New York Heart Association (NYHA) functional class (I to IV); distance covered at the six minutes walking test (metres); total hospital stay due to heart failure during 6 months before and 6 months after CRT implant (number of days).
2. Echocardiographic: LV ejection fraction (%); LV end-diastolic and end-systolic volumes (ml); presence and degree of any valvular regurgitation (from 1+ to 4+) and valvular stenosis; Doppler-derived peak pressure in pulmonary artery (mmHg); pulsed doppler pattern of transmitral flow (three types) and associated E/A ratio (abs), E wave duration (msec), A wave duration (msec), E+A waves total duration (msec).
3. Electrocardiographic: P wave, AV interval and QRS complex durations (msec); QRS axis (degrees); QRS morphology (four types: spontaneous typical or atypical left bundle branch block; RV pace-induced conduction delay; non-specific intraventricular delay).
4. Device-related: endocavitary measurements of atrial, RV and CS leads functioning (pace and sense thresholds, impedance); all programmed values of sensing and pacing; programmed AV and VV intervals; total percent time of LV pacing; burden and types of any supraventricular and ventricular tachyarrhythmias.

To define the sample size, the statistical power analysis is applied with a level of power equal to 80%, using as sample distributions the populations in the pilot study (p<0.05) and considering a drop-out rate of 20%.

Descriptive statistics are used to present and summarize the data collected in the study. For discrete variables, frequency distribution and cross tabulations are to be presented. For continuous variables, the means, standard deviations, or median and 25° and 75° percentile and ranges are used to represent data.

According to the type of variable, computed trajectory parameters are to be compared by using χ2 method, with the Fisher exact test or the nonparametric Mann-Whitney U test for non-normal distribution (p<0.05). Differences in means or in proportions are to be calculated, together with their 95% confidence intervals.

Variations in trajectory metrics from before to after pacing start are computed and correlated with variations between pre-implant and six-month post-implant assessments in both echocardiographic measures of left ventricular remodeling and function and clinical and electrocardiographic variables.

Study data are managed as follows:

* each patient is given a code to guarantee anonymity, used to identify both data on paper and imaging recordings (fluoroscopic and echocardiographic). Recordings are supplied to the Core-Labs (Bioengineering and Echocardiography) on digital support. Results from imaging recordings analyses are sent to the Principal Investigator and to the Steering Committee (composed by the Principal Investigator, the Study Directors and the Sites Principal Investigators). The original recordings are kept in each center's archives;
* all patient's data are collected on paper forms. Each center's investigator is responsible for data collection and safekeeping, and guarantees for data reliability and correctness;
* each center's data are the property of the same center; each investigator has free access to its own data and can divulge them, but without associating them with the study TRAJECTORIES. The Steering Committee alone is responsible for the whole, appropriately codified database, and can freely accede to it. Each investigator will be allowed to propose ancillary substudies/subanalyses which are to use data already provided in accordance with the protocol. Proposals have to be submitted to and approved by the Steering Committee;
* the study does not interfere with any aspect of current good clinical practice and legal requirements, and all prevailing rules will be followed.The study conforms to the guiding principles of the Declaration of Helsinki, to the current laws and to the Institutional Ethics Committee rules.The protocol has been first approved by the Area Vasta Romagna Ethics Committee, and then is submitted to other competent Ethics Committees for all participating centers;
* adverse events and adverse device effects, defined according to current standards, will be dealt with and reported to regulatory agencies and to manufacturers by each center in accordance with present regulations. The investigator ensures that, if applicable, adverse events are reported to their Ethical Committee, and/or to any Health Authorities according to national laws.

This study is conducted in accordance with Good Clinical Practice (GCP), International Standards Organization (ISO) 14155 and Declaration of Helsinki guidelines.The investigators are responsible for conducting the study in accordance with the study plan, the signed agreements, applicable laws and regulations, and any conditions of approval imposed by the reviewing Ethics Committee.

Patient informed consent is mandatory and required for all patients prior to their inclusion in the study. The process of obtaining informed consent complies with the Declaration of Helsinki and applicable national regulations, and uses language that is understandable to the patient. The informed consent form is constructed in accordance with rules given by Area Vasta Romagna Ethic Committee.The form is signed in double original, and one is given to patient, the second original kept in patients' file. The informed consent covers the use of personal information in an anonymous form and only for scientific purposes, and the acceptation of fluoroscopy as a means of clinical investigation. Patients can modify their decision at any moment, and nothing will be changed in their care and clinical programs.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent;
2. chronic systolic heart failure recognized for more than 6 months, with left ventricular systolic disfunction (ejection fraction ≤ 35%) and NYHA II-III or ambulatory IV class symptoms despite optimal medical treatment;
3. QRS complex on the surface electrocardiogram with left bundle branch block morphology and duration ≥ 120 ms, either typical or atypical or induced by right ventricular pacing due to stable chronic advanced atrio-ventricular block; QRS with with non-specific intraventricular delay lasting ≥ 150 ms;
4. a regular ventricular rhythm, either with spontaneous atrio-ventricular conduction or with ventricular pacing via a chronically implanted antibradycardia device; with sinus rhythm unless atrial fibrillation is permanent and associated with a permanent high-degree atrio-ventricular block with a spontaneous ventricular rate constantly ≤ 45 beats per minute;
5. no concomitant bradyarrhythmias being per se an indication for new implant ventricular pacing; upgrade to cardiac resynchronization therapy only if a previous pacemaker or implantable cardioverter-defibrillator was implanted more than 6 months previously;
6. a stable clinical and hemodynamic condition during cardiac resynchronization therapy device implant, and at the acquisition time heat rate between 50 and 100 beats per minute and respiratory rate ≤ 25 breaths per minute;

Exclusion Criteria:

1. inability to give informed consent;
2. occurrence of myocardial infarction, valve repair or surgery, or coronary revascularization in the past 6 months;
3. any arrhythmia at the acquisition time which frequently alters the regularity of a minimum of five consecutive heart beats;
4. participation in any other competing clinical study, with the exception of registries ruled by National Health Service Authorities or Agencies, and observational studies/registries which are not conflicting and do not interfere with any of the following aspects:

   1. the program of procedures/assessments requested by the present study;
   2. the outcome of the present study due to the requirement of medical treatments or interventions which are able to modify the clinical conditions of patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic systolic heart failure who are submitted to a cardiac resynchronization therapy device implant, with either pacemaker or implantable cardioverter-defibrillator capabilities, as a first implant or as an upgrade from a previously implanted cardiac electric device, who exhibit a normofrequent regular ventricular rhythm.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2015-01; Primary Completion 2019-01-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
the two-dimensional echocardiographic volumetric response to cardiac resynchronization therapy | six months
  the volumetric response to cardiac resynchronization therapy defined by a reduction equal or greater than 15% in two-dimensional echocardiographic end-systolic volume (ml) at six-month in comparison with pre-implant assessment;

SECONDARY OUTCOMES:
the clinical response to cardiac resynchronization therapy depicted by three metrics | six months
  the variations of three variables between pre-implant status and six-month follow-up, with no cut-off values: New York Heart Association functional class, from I to IV; distance covered at the six-minute walking test (in meters); total duration of hospital stay (number of days) due to heart failure in the 6 months before and after implant

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tomasi, M D, Principal Investigator — Ospedale Santa Maria delle Croci, Ravenna, Italy; Stefano Severi, Engeneer, Study Director — University of Bologna; Cristiana Corsi, Engeneer, Study Director — Engeneering Department , University of Bologna, Italy
Locations (7):
- Italy (7):
  - Poiliclinico Sant'Orsola-Malpighi, Bologna, BO
  - Ospedale Maurizio Bufalini, Cesena, FC
  - Ospedale Santa Maria delle Croci, Ravenna, RA
  - Ospedale Mater Salutis, Legnago, Verona
  - Ospedale Classificato Equiparato Sacro Cuore - Don Calabria -, Negrar, VR
  - Ospedale S Maria della Misericordia - AUSL 18 del Veneto, Rovigo
  - Ospedale San Bortolo, Vicenza